CLINICAL TRIAL: NCT05349578
Title: A Prospective Comparison of Cotton Swab Method and Conventional Biopsy Sampling in Rapid Urease Test for Helicobacter Pylori Detection
Brief Title: Gastric Swab for Helicobacter Pylori Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyunsoo Chung, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2108-016-1247
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; rapid urease test; swab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue (Other): conventional RUT using biopsied tissue
  Interventions: Diagnostic Test: swab RUT
- Swab (Experimental): RUT using swab
  Interventions: Diagnostic Test: swab RUT

INTERVENTIONS:
Diagnostic Test: swab RUT — rapid urease test using swab instead of biopsied tissue

SUMMARY:
A randomized controlled trial for comparing the Helicobacter pylori test using the swap method and the method using the conventional biopsy.

DETAILED DESCRIPTION:
The aim of this study is to conduct a prospective study under the hypothesis that a cotton swab method in the rapid urease test is not inferior to the conventional biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-80
* Patients who undergo esophagogastroduodenoscopy and need for investigation of Helicobacter pylori infection.

Exclusion Criteria:

* Surgical history of any kind of gastrectomy
* Patients with contraindication of esophagogastroduodenoscopy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Accuracy | the same day wtih EGD
  Accuracy of diagnosis for Helicobacter pylori infection

SECONDARY OUTCOMES:
sensitivity, false positive, false negative rate, etc. | the same day wtih EGD

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soh H, Kim N, Moon J, Lee HM, Kim B, Cho SJ, Kim SG, Chung H. Gastric mucosal swab as an alternative to biopsy for Helicobacter pylori detection. Helicobacter. 2023 Jun;28(3):e12980. doi: 10.1111/hel.12980. Epub 2023 Apr 7. PMID 37026561